CLINICAL TRIAL: NCT02339493
Title: Alert-Based Computerized Decision Support for Stroke Prevention in High-Risk Hospitalized Patients With Atrial Fibrillation: A Randomized, Controlled Trial (AF-ALERT)
Brief Title: Electronic Alerts for Stroke Prevention in Patients With Atrial Fibrillation or Atrial Flutter
Acronym: AF-ALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Samuel Z.Goldhaber, MD, Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014P002317
Record Dates: First submitted 2015-01-06; First posted 2015-01-15 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alert Group (Experimental): If the patient is randomized to the alert group, their ordering provider will receive a computer electronic alert notifying the responsible provider that his or her patient is high-risk for stroke due to AF or atrial flutter and that the patient is not ordered to receive anticoagulant therapy.
  Interventions: Other: Computer Electronic Alert
- Control Group (No Intervention): If the patient is randomized to the control group, the computer program will not issue an on-screen electronic alert.

INTERVENTIONS:
Other: Computer Electronic Alert — A computer program that will issue an on-screen electronic alert notifying the responsible provider that his or her patient is high-risk for stroke due to AF or atrial flutter and that the patient is not ordered to receive anticoagulant therapy. The alert will provide options for anticoagulation for stroke prevention in AF as well as additional information in the form of suggested reading.
  Arms: Alert Group

SUMMARY:
Atrial fibrillation (AF) is the most preventable cause of stroke. CHADS and CHA2DS2VASc scores predict the likelihood of stroke in patients with nonvalvular AF. Atrial flutter confers a similar risk of stroke as atrial fibrillation. Anticoagulant therapy with warfarin, dabigatran, rivaroxaban, apixaban, and edoxaban is effective for prevention of thromboembolic stroke in most patients with AF. However, despite widely available risk stratification tools, five options for anticoagulation, and evidence-based practice guidelines, thromboprophylaxis for stroke prevention in AF is under-prescribed in the U.S., Europe, and worldwide. The investigators have previously demonstrated the efficacy of an alert-based computerized decision support (CDS) strategy for prevention of symptomatic venous thromboembolism (VTE) in at-risk hospitalized patients not receiving any thromboprophylaxis. The investigators' goal is to create and evaluate an alert-based CDS strategy for stroke prevention in patients with nonvalvular AF or atrial flutter in a randomized controlled trial.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most preventable cause of stroke. CHADS and CHA2DS2VASc scores predict the likelihood of stroke in patients with nonvalvular AF. Atrial flutter confers a similar risk of stroke as atrial fibrillation. Anticoagulant therapy with warfarin, dabigatran, rivaroxaban, apixaban, and edoxaban is effective for prevention of thromboembolic stroke in most patients with AF. However, despite widely available risk stratification tools, five options for anticoagulation, and evidence-based practice guidelines, thromboprophylaxis for stroke prevention in AF is under-prescribed in the U.S., Europe, and worldwide. The investigators have previously demonstrated the efficacy of an alert-based computerized decision support (CDS) strategy for prevention of symptomatic venous thromboembolism (VTE) in at-risk hospitalized patients not receiving any thromboprophylaxis. The investigators' goal is to create and evaluate an alert-based CDS strategy for stroke prevention in patients with nonvalvular AF or atrial flutter in a randomized controlled trial. The investigators have the following specific aims:

Aim #1 (Primary Efficacy Endpoint)- To assess whether an alert-based computerized decision support strategy increases prescription of anticoagulation during hospitalization, at discharge, and at 90 days from enrollment.

Hypothesis #1- An alert-based computer decision support (CDS) strategy will increase prescription of prescription of anticoagulation during hospitalization, at discharge, and at 90 days from enrollment.

Aim #2 (Secondary Efficacy Endpoint)- To determine the potential impact of an alert-based computerized decision support strategy on the frequency of a composite of major adverse cardiovascular events at 90 days, defined as cerebrovascular accident, systemic embolism, myocardial infarction (MI), and all-cause mortality at 90 days from enrollment.

Hypothesis #2- This study will provide proof-of-concept data, including event rates, from which to design a larger randomized control trial to assess whether an alert-based CDS strategy will reduce the frequency of a composite of major adverse cardiovascular events at 90 days, defined as cerebrovascular accident, systemic embolism, myocardial infarction (MI), and all-cause mortality at 90 days from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients ≥ 21 years old with paroxysmal, persistent, or permanent nonvalvular AF or atrial flutter (CHA2DS2VASc score ≥ 1) who are not prescribed anticoagulant therapy for stroke prevention and are hospitalized at BWH will be eligible for randomization.

Exclusion Criteria:

* <21 years old
* no diagnosis of AF or atrial flutter
* not hospitalized at BWH

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Frequency of prescription of anticoagulation during hospitalization, at discharge, and at 90 days from enrollment. | 90 days
  Defined as prescription of therapeutic dose anticoagulation

SECONDARY OUTCOMES:
Frequency of composite of major adverse cardiovascular events at 90 days | 90 days
  Defined as cerebrovascular accident, systemic embolism, myocardial infarction (MI), and all-cause mortality at 90 days from enrollment
Frequency of stroke or transient ischemic attack (TIA) at 90 days | 90 days
  An acute stroke was defined as a new, focal neurologic deficit of sudden onset, lasting at least 24 hours, not due to a readily identifiable nonvascular cause (e.g., brain tumor, trauma), as confirmed by a neurologist. All strokes required confirmation by imaging or autopsy. TIA was defined as a transient episode of neurologic dysfunction caused by suspected focal cerebral, spinal cord, or retinal ischemia without evidence of acute infarction and confirmed by a neurologist.
Frequency of acute myocardial infarction at 90 days | 90 days
  Acute MI was defined as the detection of a rise and/or fall of cardiac biomarkers (cardiac troponin T), with at least one value being elevated above the 99th percentile upper reference limit and with at least one of the following: 1) symptoms of myocardial ischemia; 2) new (or presumably new) significant ST-segment/T-wave changes or left bundle branch block; 3) development of pathological Q waves on ECG; 4) new loss of viable myocardium or regional wall motion abnormality by imaging; or 5) identification of intracoronary thrombus by angiography or autopsy.
Frequency of all cause mortality at 90 days | 90 days
  All-cause mortality was determined by review of the EHR. Causes of death were classified as stroke, myocardial infarction, pulmonary embolism, other cardiovascular cause, bleeding, cancer, or non-cardiovascular and non-cancer.
Frequency of major bleeding or clinically relevant non-major bleeding at 90 days | 90 days
  Defined by the International Society on Thrombosis and Haemostasis [ISTH] bleeding classification system) at 90 days from enrollment.14 Using the ISTH classification, bleeding was defined as major if it was overt and associated with a decrease in the hemoglobin level of 2 g/dL or more, required the transfusion of 2 or more units of blood, occurred into a critical site, or contributed to death. Clinically relevant non-major bleeding was defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, surgical intervention, or interruption of the study drug.
Frequency of systemic embolism at 90 days | 90 days
  Systemic embolism was defined as sudden loss of perfusion of a limb or extracranial organ

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piazza G, Hurwitz S, Carroll B, Goldhaber SZ. Patients with perceived high-bleeding risk and computerized decision support for stroke prevention in atrial fibrillation: an AF-ALERT substudy : Piazza: outcomes of high-bleeding risk AF patients. J Thromb Thrombolysis. 2021 Jul;52(1):281-290. doi: 10.1007/s11239-020-02296-0. Epub 2020 Sep 30. PMID 33000390
- [Derived] Piazza G, Hurwitz S, Galvin CE, Harrigan L, Baklla S, Hohlfelder B, Carroll B, Landman AB, Emani S, Goldhaber SZ. Alert-based computerized decision support for high-risk hospitalized patients with atrial fibrillation not prescribed anticoagulation: a randomized, controlled trial (AF-ALERT). Eur Heart J. 2020 Mar 7;41(10):1086-1096. doi: 10.1093/eurheartj/ehz385. PMID 31228189